CLINICAL TRIAL: NCT03799601
Title: A Single Arm, Multi-center Study to Assess the Efficacy and Safety of Docetaxel Combined With Carboplatin Plus Anlotinib as First Line Treatment in Non-squamous Non-small-cell Lung Cancer (NSCLC)
Brief Title: Docetaxel Combined With Carboplatin Plus Anlotinib as First Line Treatment in NSCLC
Acronym: ALTER-L013
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJCC-LC-20190108
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: NSCLC
Keywords: Anlotinib; Docetaxel; Carboplatin; NSCLC
MeSH Terms: interventions — anlotinib; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination of docetaxel, carboplatin and anlotinib (Experimental)
  Interventions: Drug: Anlotinib; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Anlotinib — Anlotinib which has shown an affirmatory efficacy in ALTER0303 controlled trial as a 3rd-line treatment on advanced NSCLC is a tyrosine kinase inhibitor with a favorable safety profile in phase I trial which mainly targets VEGFR1/2/3, FGFR, PDGFR and c-kit.
  Other Names: Anlotinib Hydrochloride
Drug: Docetaxel — a chemotherapy medication used to treat a number of types of cancer.This includes breast cancer, head and neck cancer, stomach cancer, prostate cancer and non-small-cell lung cancer.It may be used by itself or along with other chemotherapy medication.It is given by slow injection into a vein.
Drug: Carboplatin — Carboplatin is used to treat a number of forms of cancer. This includes ovarian cancer, lung cancer, head and neck cancer, brain cancer, and neuroblastoma. It may be used for some types of testicular cancer but cisplatin is generally more effective.

SUMMARY:
Anlotinib which has shown an affirmatory efficacy in ALTER0303 controlled trial as a 3rd-line treatment on advanced NSCLC is a tyrosine kinase inhibitor with a favorable safety profile in phase I trial which mainly targets VEGFR1/2/3, FGFR, PDGFR and c-kit. The purpose of this trail is to establish whether advanced non-squamous NSCLC patients could benefit from the combination treatment of docetaxel, carboplatin and anlotinib as the first-line and maintenance treatment.

DETAILED DESCRIPTION:
First-line patients (or postoperative recurrence) with locally advanced or metastatic NSCLC were enrolled in this trail. The patients (clinical stage ⅢB/Ⅳ, with no sensitizing mutation of the epidermal growth factor receptor gene or translocation of the anaplastic lymphoma kinase gene) were confirmed by histological or cytological diagnosis. The primary endpoint is PFS; secondary endpoint includes OS, DCR and ORR. The study was single-arm, conducted at 8 centers in China mainland. The primary end point was PFS (time from enrollment to first RECIST1.1-defined PD or death). 45 patients were planned for enrollment. This estimate was based on 80% power, with a two-sided 5% significance level. We analyzed PFS and OS using Kaplan-Meier methodology. The research protocol was approved by the relevant ethics committees, and the study was conducted according to the Declaration of Helsinki and Good Clinical Practice guidelines. Patients gave written informed consent to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age on the day of signing informed consent and with good compliance and agree to accept follow-up of disease progression and adverse events.
* Patients with histologic or cytologic confirmation of advanced or metastatic Non squamous NSCLC with stage IIIB or IV disease.（For recurrent patients, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant were assessed for eligibility, and the last treatment time must be more than 6 months before enrollment）
* There were at least one target lesions in the past three months has not yet accepted radiotherapy, and could be recorded by magnetic resonance imaging (MRI) or computer tomography (CT) measuring accurately at least in one direction(The maximum diameter needs to be recorded), including conventional CT ≥20 mm or spiral CT ≥10 mm.
* Life expectancy ≥6 months
* a performance status of 0 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* With normal marrow, liver ,renal and coagulation function:
* The blood routine examination need to be standard (no blood transfusion and blood products within 14 days, no g-csf and other hematopoietic stimulating factor correction)
* The main organs function are normally, the following criteria are met:(1)Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimuli): HB≥90 g/L; ANC ≥ 1.5×10^9/L; PLT ≥80×10^9/L;(2)Biochemical examinations must meet the following criteria: TBIL<1.5×ULN; ALT and AST < 2.5×ULN, and for patients with liver metastases < 5×ULN; Serum Cr ≤ 1.25×ULN or endogenous creatinine clearance > 60 ml/min (Cockcroft-Gault formula);
* Women of child-bearing age should take appropriate contraceptive measures and should not breastfeed from screening to 3 months after stopping the study and treatment.Before starting administration, the pregnancy test was negative, or one of the following criteria was met to prove that there was no risk of pregnancy:

  1. Postmenopause is defined as amenorrhea at least 12 months after age 50 and cessation of all exogenous hormone replacement therapy;
  2. Postmenopausal women under the age of 50 May also be considered postmenopausal if their amenorrhea is 12 months or more after the cessation of all exogenous hormone therapy and their luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the reference value range of laboratory postmenopausal;
  3. Have undergone irreversible sterilization surgery, including hysterectomy, bilateral ovectomy or bilateral salpingectomy, except for bilateral tubal ligation.
* For men, consent is required to use appropriate methods of contraception or to be surgically sterilized during the trial and 8 weeks after the last administration of the trial drug.

Exclusion Criteria:

* Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer), Lung sarcomatoid carcinoma;
* Had histologically confirmed lung squamous cell carcinoma, or adenosquamous carcinoma;
* Patients with pathological fracture in bone metastasis induced by non-small-cell lung cancer;
* Tumor histology or cytology confirmed EGFR mutagenesis [EGFR sensitive mutations include 18 exon point mutations (G719X), 19 exon deletions, 20 exon S768I mutations and 21 exon point mutations (L858R and L861Q)] and ALK gene rearrangement positivity, include EGFR/ALK status cannot be determined for various reasons;
* Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor; Medical history and combined history：
* Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 28 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms and metastases in midbrain, pons, cerebellum, medulla oblongata, or spinal cord, brain metastases and local radiotherapy after two weeks to allow group);
* The patient is participating in other clinical studies or completing the previous clinical study in less than 4 weeks;
* Had malignant tumors except NSCLC within 5 years before enrollment(except for patients with carcinoma in situ of the cervix , basal cell or squamous cell skin cancer who have undergone a curative treatment, local prostate cancer after radical resection, ductal carcinoma in situ or papillary thyroid cancer after radical resection);
* Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy; Note: Under the condition of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes;
* Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
* The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma;
* Severe acute or chronic infections requiring systemic treatment; Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
* There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
* Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment; Long-term unhealed wounds or fractures;
* Decompensated diabetes or other ailments treated with high doses of glucocorticoids;
* Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
* Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
* Events of venous/venous thrombosis occurring within the first 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Physical examination and laboratory findings:

  1. A known history of HIV testing positive or acquired immunodeficiency syndrome (AIDS);
  2. Untreated active hepatitis (hepatitis b: HBsAg positive and HBV DNA more than 1 x 103 copy /ml; Hepatitis c: HCV RNA is positive and liver function is abnormal); Combined with hepatitis b and hepatitis c infection;
  3. Serious diseases that endanger patients' safety or affect patients' completion of research,according to the researchers' judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | Estimated about 24 months.
  Clinical response of treatment according to RESIST v1.1 criteria (PFS, progression-free survival)

SECONDARY OUTCOMES:
Overall Survival | Estimated about 24 months.
  Clinical response of treatment according to RESIST v1.1 criteria (OS, overall survival)
Disease Control Rate | Estimated about 24 months.
  Clinical response of treatment according to RESIST v1.1 criteria (DCR, disease control rate)
Overall Response Rate | Estimated about 24 months.
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, Overall Response Rate)

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology,, Wuhan, Hubei, China